CLINICAL TRIAL: NCT06969144
Title: Subtotal Cholecystectomy for Difficult Gall Bladder Due to Chronic Cholecystitis: A Cross-sectional Study
Brief Title: Subtotal Cholecystectomy for Difficult Gall Bladder Due to Chronic Cholecystitis
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Ishwor Thapaliya, Principal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 416(6-11)E2,081/82
Record Dates: First submitted 2025-01-27; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-01

CONDITIONS: Gallstone
MeSH Terms: conditions — Gallstones | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | US Export: No

INTERVENTIONS:
Procedure: cholecystectomy — The indications for elective cholecystectomy were symptomatic cholelithiasis, a GB polyp more than ten millimeters, a history of cholecystitis, biliary pancreatitis, or choledocholithiasis. Patients with cholecystitis and severe or moderately severe pancreatitis were operated on after six weeks of the event. Other patients received surgery at the earliest available date. All patients with choledocholithiasis underwent endoscopic retrograde cholangiopancreatography (ERCP) and stone clearance before cholecystectomy. Patients who underwent laparoscopic cholecystectomy were evaluated by surgical and anesthesia teams in outpatient clinics and co-morbid conditions were optimized. Preoperative antibiotic prophylaxis was given to all the patients before induction of anesthesia.

SUMMARY:
Subtotal cholecystectomy (STC) is a valuable technique when severe inflammation, fibrosis, or anatomical variations obscure the critical view of safety essential for identifying the cystic duct and artery. It helps reduce the risk of bile duct injuries and other complications that arise during a total cholecystectomy (TC) when these structures are not visible. This study evaluates the safety and outcomes of subtotal cholecystectomy in chronic cholecystitis.

DETAILED DESCRIPTION:
A retrospective analysis was conducted in all patients who underwent a cholecystectomy between May 2021 and November 2024. Indications, complications, and perioperative outcomes of STC were compared with those of standard TC.

The investigators concluded STC is an important bailout procedure in a difficult laparoscopic cholecystectomy associated with higher early postoperative complications but lower bile duct injury.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cholelithiasis planned for laparoscopic cholecystectomy
* Clinical diagnosis of gallbladder polyp planned for laparoscopic cholecystectomy

Exclusion Criteria:

* Gall bladder malignancy
* Cholelithiasis and gallbladder polyp cases managed non-operatively
* additional procedures along with cholecystectomy like bile duct exploration, bile duct excision for choledochal cyst.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 1149 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
postoperative outcomes of subtotal cholecystectomy (STC) and total cholecystectomy (TC) | upto 22 months
  The primary outcome was to assess the postoperative outcomes of subtotal cholecystectomy (STC) and total cholecystectomy (TC) groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Nepal, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
apart from identifiers, relevant clinical data.
Supporting Information: Study Protocol, ICF
Time Frame: as supplementary file
Access Criteria: as supplementary file